CLINICAL TRIAL: NCT07118267
Title: The Intervention of Lactobacillus Plantarum Probiotics in Adult Patients With Autistic Spectrum Disorders Investigating Associations of Microbiota, Inflammation, Social Interactions, Quality of Life, and Gait Analysis: A Qualitative and Quantitative Mixed & A Double-blind Randomized Controlled Trial
Brief Title: The Intervention of Lactobacillus Plantarum Probiotics in Adult Autistic Spectrum Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Shu-I Wu, Attending Physician, Mackay Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24MMHIS529e; 114-2314-B-195-015- (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Autism Disorder
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- probiotics (Experimental): Lactobacillus plantarum
  Interventions: Dietary Supplement: Lactiplantibacillus plantarum

INTERVENTIONS:
Dietary Supplement: Lactiplantibacillus plantarum — containing 60 billion CFU (administered as two capsules per day)

SUMMARY:
This is a qualitative and quantitative mixed-methods, open-label study, will involve 12 participants and their caregivers. Participants will also undergo blood exams and gait analysis, while caregivers will complete qualitative interviews and quantitative questionnaires on autistic symptoms, stress, anxiety, and quality of life. After the baseline assessments, participants will receive Lactobacillus plantarum for 8 weeks, followed by further evaluations at end point.

DETAILED DESCRIPTION:
One neurodevelopmental disease that manifests before the age of three is autism. It is a range of widespread developmental problems that affect people from various socioeconomic backgrounds and ethnicities. Beginning in 2013, autism spectrum disorder (ASD) becomes the general diagnosis given to all children with autism, Asperger's syndrome, or other prevalent developmental abnormalities (DSM-5, APA). Over the past two decades, the frequency of ASD has steadily increased. Greater awareness of the problem or easier access to diagnostic services could be the cause of this.

Children with ASD have difficulties in social interaction, communication, and language skills with many children demonstrating delayed language development, unusual speech patterns, lack of spoken language, challenges in forming peer relationships, restrictive and repetitive behaviours such as rocking or hand flapping, or over- or under-reactive to stimuli. In adults with ASD, they may still have blunt or literal communication style, preference for solitude, difficulty understanding social cues, challenges in maintaining conversations, discomfort in social situations, adherence to routines, repetitive behaviors and sensory sensitivities similar to those seen in childhood but probably more controlled or masked. While the core characteristics of ASD remain consistent, the manifestation of symptoms can change with age and development. Talking with caregivers and other family members to find out about the person's early developmental history will help ensure an accurate diagnosis when diagnosing and evaluating people with ASD. Many adults with ASD struggle with finding and keeping employment, which can affect their independence and quality of life. ASD adults may also have co-occurring health conditions, such as anxiety and depression, which further impact daily functioning and overall well-being.

In recent years, the microbiota and the gut-brain axis (MGB, or the biochemical signaling pathway that connects the gastrointestinal tract and the nervous system) has attracted much attention in regulations and interactions of the nervous and immune systems. Intestinal microbes and their metabolites have been shown to regulate the human body through a series of biochemical and functional linkages. The microbiota is considered to be an essential organ of the human body for maintaining homeostasis. The composition of the intestinal flora is not only related to factors such as age, diet, or metabolic diseases, but also plays key roles in absorption, storage, metabolism, and maintenance of healthy immune function.

As for human research, Proteobacteria, Firmicutes, and Bacteroides are the three primary types of microorganisms found in the gut. They must be in harmony with one another; in fact, dysbiosis, an imbalance, can have an impact on gut health. Recent studies have started to investigate associations of microbiota and mental disorders, including depression or anxiety, autistic spectrum disorder, schizophrenia, or bipolar disorder.

ASD has primarily been examined in clinical trials conducted on children to examine the impacts of probiotics on neurological disorders. The main clinical trials on the effects of probiotics on children with ASD showed both the benefits and the drawbacks. Different probiotic dosages and results employing various beneficial microorganisms have been reported in trials looking into probiotic therapy in children with ASD.

While there's a growing body of research suggesting a potential link between gut health and neurodevelopmental disorders like ASD, most clinical trials of probiotics have been focusing on children. As of now, there aren't many large-scale, randomized controlled trials specifically targeting adults with ASD and probiotic interventions. However, the increasing recognition of the gut-brain axis and the potential benefits of probiotics in various conditions, including mental health, makes this an area of active research. The gut microbiome and its influence on brain function may differ between children and adults. The long-term effects of probiotic interventions on adult ASD symptoms need to be evaluated. The response to probiotic therapy can vary significantly among individuals due to the complex nature of ASD. While there's promising potential, more rigorous scientific research is required to establish the efficacy and safety of probiotics as a treatment for adults with ASD. However, research on the effects of probiotics or Lactobacillus plantarum on adults with ASD diagnosed in childhood still lacking. This study aims to examine whether Lactobacillus plantarum may be a possible new dietary approach for improving behavioral symptoms and enhancing the quality of life of caregivers among adults ASD diagnosed since childhood. This study also intends to outline the potential mechanisms by which the probiotics' direct or mediating effects can alleviate the microbiota-gut-grain dysfunction in the management of adults with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with autistic spectrum disorder aged 18~50 years old
* Those whose primary contacts or caregiver (including family members or teachers) are willing to participate
* Those whose primary contacts or caregivers can understand Mandarin and can answer relevant questions or questionnaires.

Exclusion Criteria:

* Have taken antibiotics or are receiving antibiotic treatment within one month.
* Have used probiotic products in powder, capsule or tablet form within two weeks (excluding yogurt, Yakult and other related foods).
* Patients who have undergone hepatobiliary gastrointestinal surgery (except for colorectal polypectomy and appendectomy).
* Past or current patients with inflammatory bowel disease.
* Those with a history of cancer.
* Those who are allergic to lactic acid bacteria products.
* Those who are receiving parenteral nutrition.
* Those who are evaluated by the principal investigator to be unsuitable to participate in the research.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Clinical Global Impression of Improvement (CGI-I) | baseline to week8
  Patient Clinical Global Impression of Improvement (CGI-I) scale rated by the patient is a 7-point scale of improvement from 'very much improved' to 'very much worse'. 'Very much improved' means a better outcome.

SECONDARY OUTCOMES:
The Autism Behavior Checklist-Taiwan, ABCT | baseline to week 8
  The Checklist scale contains 47 items: 8 items pertaining to sensory (sensation and perception), 11 items to relating (social connection), 12 items pertaining to body and object use (motor activity and rigid object use), 8 items pertaining to language (communication and interaction), and 8 items pertaining to social and self-Help (adaptability and self-care). The scoring method gives 1 point for each "Yes" answer. The higher the score, the more severe the autistic behaviors. This scale has favorable content consistency, with a Cronbach α value between 0.75 and 0.87, retest reliability at 0.89. The content validity and reliability of the scale are satisfactory.
Parent Target Symptom Rating Visual Analogue Scale, PTSVAS | baseline to week 8
  A 100mm horizontal scale will be used to evaluate the descriptions and ratings, with each 10mm segment representing one unit. The scale ranges from "very good" or "completely resolved" (0) to "worst" or "catastrophic worsening" (10), with 5 representing no change.
Parenting Stress Index Fourth Edition Short Form, PSI-4-SF | baseline to week 8
  The PSI-4-SF yields scores on the following subscales: 1) Parental Distress, 2) Parent-Child Dysfunctional Interaction, and 3) Difficult Child. The instrument has 36 items which are responded to on a 5-point scale ranging from Strongly Agree to Strongly Disagree. A Total Stress Score is obtained by combining the subscales. The software to score the PSI-4-SF provides a percentile score. Percentile scores between 16 and 84% are considered normal stress, while scores of 85-89% indicate high stress and scores of 90% or higher indicate stress levels that may be clinically significant.
Quality of Life in Autism Questionnaire, QoLA | baseline to week 8
  The "Quality of Life in Autism Questionnaire" (QoLA) is a scale specifically designed for parents or caregivers of children with autism, aiming to assess their quality of life. The questionnaire consists of two parts:
  Part A: Evaluates the overall sense of quality of life experienced by the parent or caregiver. This section includes various items such as: "I feel happy and content" and "I am satisfied with my social life." Part B: Assesses the impact of the child's autism symptoms or characteristics on the parent or caregiver. The items in this section aim to understand how the child's autistic traits affect family life and the parent's daily experiences.
  The full questionnaire contains 48 items and is designed to comprehensively evaluate both the quality of life of the parent or caregiver and the impact of the child's autism symptoms on them.

CONTACTS AND LOCATIONS:
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided